CLINICAL TRIAL: NCT00084825
Title: Crossover From Docetaxel and Placebo to Docetaxel and Imatinib in Patients With Androgen-Independent Prostate Cancer With Bone Metastases: Extension Trial to ID03-0008
Brief Title: Docetaxel and Imatinib Mesylate in Treating Patients With Androgen-Independent Prostate Cancer and Bone Metastases That Progressed on the Docetaxel and Placebo Group of MDA-ID-030008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000365625; MDA-ID-030222; MSKCC-03149; ID03-0222 (Other: UT MD Anderson Cancer Center)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Docetaxel; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel + Imatinib Mesylate (Experimental): Docetaxel intravenous (IV) over 1 hour on days 1, 8, 15, and 22 and oral imatinib mesylate once daily on days 1-42. Courses repeat every 42 days.
  Interventions: Drug: Docetaxel; Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Docetaxel — 30 mg/m^2 IV on days 1, 8, 15, and 22 every 42 days
Drug: Imatinib mesylate — 600 mg orally daily

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as docetaxel work in different ways to stop tumor cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving docetaxel with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel with imatinib mesylate works in treating patients with androgen-independent prostate cancer and bone metastases that progressed while receiving docetaxel and a placebo on clinical trial MDA-ID-030008.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Provide treatment with docetaxel and imatinib mesylate for patients with androgen-independent prostate cancer and bone metastases that progressed while receiving docetaxel and placebo on MDA-ID-030008.

Secondary

* Determine the response rate and time to progression in these patients after crossover from docetaxel and placebo to docetaxel and imatinib mesylate.
* Compare the modulation of the platelet-derived growth factor receptor pathway by docetaxel and imatinib mesylate vs docetaxel and placebo in the same patient.
* Determine the quality of life of patients treated with this crossover regimen.

OUTLINE: This is an open-label, crossover, multicenter, extension study. Patients who progressed on the placebo and docetaxel arm of MDA-ID-030008 crossover to receive docetaxel and imatinib mesylate.

Patients receive docetaxel IV over 1 hour on days 1, 8, 15, and 22 and oral imatinib mesylate once daily on days 1-42. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each therapy course, and at the completion of therapy.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A maximum of 72 patients will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Osseous metastases
* Androgen-independent disease
* Previously randomized to the docetaxel and placebo arm of protocol MDA-ID-030008 and has been removed from protocol due to disease progression

  * No more than 6 weeks since final treatment with docetaxel and placebo
* No uncontrolled brain metastases or spinal cord compression

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-3

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 2 times upper limit of normal
* No chronic liver disease

Renal

* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* No New York Heart Association class III or IV congestive heart failure
* No unstable angina
* No uncontrolled severe hypertension
* No myocardial infarction within the past 6 months

Pulmonary

* No oxygen-dependent lung disease

Other

* No prior dose-limiting toxicity with docetaxel requiring more than 2 dose reductions
* No severe hypersensitivity to docetaxel
* No prior dose-limiting toxicity with docetaxel requiring 1 dose reduction AND experienced recurrent grade 3 or 4 toxicity at the time of progression on MDA-ID-030008
* No uncontrolled diabetes mellitus
* No concurrent severe infection
* No overt psychosis, mental disability, or other incompetency that would preclude giving informed consent
* No history of non-compliance
* HIV negative
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent second-line hormonal therapy

Radiotherapy

* At least 3 weeks since prior radiotherapy
* No recent strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium

Surgery

* Recovered from prior surgery

Other

* No other concurrent anticancer agents
* No other concurrent investigational agents
* No concurrent therapeutic warfarin

  * Concurrent mini-dose warfarin (1 mg/day) for central venous catheter prophylaxis allowed
* No concurrent grapefruit or grapefruit juice

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-05; Primary Completion 2006-07 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy | 12 weeks after initiation of crossover therapy

SECONDARY OUTCOMES:
Time to progression | From registration to disease progression, up to 32 months
  Time of progression was defined as the time of appearance of symptoms attributable to disease progression, the first demonstrated clinical sign or radiological evidence of disease progression, or the time of first of consecutive prostate-specific antigen (PSA) increments that achieved 25% increase over baseline or nadir (or death during the study), whichever was earliest.
Response rate | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, Study Chair — M.D. Anderson Cancer Center; Christopher Logothetis, MD, Study Chair — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Result] Mathew P, Thall PF, Johnson MM, et al.: Preliminary results of a randomized placebo-controlled double-blind trial of weekly docetaxel combined with imatinib in men with metastatic androgen-independent prostate cancer (AIPC) and bone metastases (BM). [Abstract] J Clin Oncol 24 (Suppl 18): A-4562, 232s, 2006.
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org